CLINICAL TRIAL: NCT06710223
Title: A Phase Ib Study of Cryoablation and Pressure-enabled Hepatic Arterial Infusion of Class C Toll-like Receptor 9 Agonist SD-101 in Combination with Durvalumab and Tremelimumab in Patients with Advanced Hepatocellular Carcinoma
Brief Title: Cryoablation and Arterial Infusion of SD-101 in Combination with Durvalumab and Tremelimumab
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Principal Investigator, Adam Burgoyne, MD, PhD, Associate Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810313
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cryotherapy; tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SD-101 (Experimental): Participants will be treated with cryoablation and intrahepatic artery infusion of SD-101. This treatment will be followed by administration of the immune checkpoint inhibitors Tremelimumab and Durvalumab (STRIDE regimen). Tremelimumab 300mg will be given intravenously once, 7-10 days after cryoablation + SD-101. Durvalumab 1500mg will be given intravenously at the same time as Tremelimumab, and then every 28 days (on day 1 of every subsequent cycle).
  Interventions: Drug: SD-101; Device: Cryotherapy; Drug: Tremelimumab; Drug: Durvalumab

INTERVENTIONS:
Drug: SD-101 — Toll-like receptor 9 (TLR9) agonist
  Other Names: nelitolimod
Device: Cryotherapy — Cryoablation of liver
Drug: Tremelimumab — Anti-CTLA4
Drug: Durvalumab — Anti-PDL1

SUMMARY:
The goal of this Phase 1b clinical trial is to evaluate the safety and efficacy of cryoablation and hepatic arterial administration of SD-101 in participants with advanced hepatocellular carcinoma. After this procedure, participants will be treated with tremelimumab and durvalumab every 4 weeks (STRIDE regimen).

DETAILED DESCRIPTION:
This is a phase I, single site study to determine the safety, tolerability, and efficacy of cryoablation combined with hepatic arterial administration of SD-101 in participants with advanced hepatocellular carcinoma (HCC). After this procedure, participants will be treated with tremelimumab and durvalumab every 4 weeks (STRIDE regimen).

SD-101 (also called nelitolimod) is a CpG oligodeoxynucleotide (CpG-ODN). More specifically, SD-101 is a bacterial DNA fragment that functions as a toll-like-receptor 9 (TLR9) agonist on myeloid-derived suppressor cells (MDSC), plasmacytoid dendritic cells (pDC), and other immune cells. TLR9 activation by SD-101 reprograms the tumor microenvironment (TME) and activates the immune system, rendering the tumor more susceptible to cancer immunotherapies, such as immune checkpoint inhibitors (ICI).

This study will administer SD-101 by pressure-enabled drug delivery (PEDD) directly into the hepatic artery during the tumor cryoablation procedure. This treatment will be followed by the STRIDE regimen, which consists of the administration of 2 immune checkpoint inhibitors: single dose of the anti-Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) antibody tremelimumab at 300 mg and once-monthly dose of the anti-Programmed Death-Ligand 1 (PDL1) antibody durvalumab at 1500 mg.

The hypothesis of this phase I study is that treatment with SD-101 will improve the efficacy of tremelimumab plus durvalumab by stimulating a robust systemic antitumoral immune response.

Patients with advanced HCC eligible for ICI treatment will be enrolled. Seven to ten days before the first ICI dose, participants will undergo ultrasound- and/or CT-guided cryoablation of part of a single hepatic lesion and concurrent administration of SD-101. US-guided liver biopsy will also be performed immediately prior to cryoablation as well as 30 days (plus or minus 7 days) afterwards. Participants will continue on ICI therapy infusions per the STRIDE regimen and tumor response will be evaluated by contrast-enhanced multiphase MRI or CT every 8 weeks (plus or minus 7 days) for 1 year. After the first year, tumor assessment will be conducted every 12 weeks (plus or minus 14 days).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to performance of any study- specific procedures.
* Age ≥ 18 years.
* Locally advanced or metastatic and/or unresectable hepatocellular carcinoma (HCC) with diagnosis confirmed by histology/cytology or clinically by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic participants:

  1. For cirrhotic participants with no histological confirmation of diagnosis, clinical confirmation is required per AASLD criteria.
  2. Pathological diagnoses of HCC will be made according to the International Working Party criteria.
* HCC with a component that measures at least 3 cm and that is located 1 cm or greater away from sensitive structures, including large blood vessels, large bile ducts, pericardium, diaphragm, gallbladder, stomach, and bowel.
* Is not a candidate for local therapies alone, including liver transplantation, tumor ablation, transarterial embolization, radiation therapy, or resection.
* No prior systemic therapy for advanced or metastatic HCC.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Evaluable target lesions as per Response Evaluation Criteria in Solid Tumors RECIST v1.1 or mRECIST.
* Child-Pugh A or Child-Pugh B7 liver function.
* Life expectancy of ≥ 12 weeks.
* Adequate bone marrow function defined as:

  1. Peripheral absolute neutrophil count ≥ 1000/mm^3
  2. Platelet count ≥ 50,000/ mm^3
  3. Hemoglobin ≥ 8.0 g/dL
* Adequate renal function defined as creatinine clearance ≥ 50 ml/min
* Adequate liver and pancreatic function defined as:

  1. Total bilirubin ≤ 2.0 x institution's upper limit of normal, and
  2. Alanine transaminase (ALT) or Aspartate transaminase (AST) ≤ 5 x institution's upper limit of normal, and
  3. Albumin ≥ 2 g/dL
* Adequate central nervous system function defined as:

  a. patients with seizure disorder may be enrolled if on anticonvulsants and seizures are well controlled.
* Systolic blood pressure <160 mm Hg.
* Patients with partners of childbearing potential must agree to use adequate contraception during participation in the study.
* Patients able to become pregnant are eligible to enter the study if they are either:

  1. Of non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including: i. Has had a hysterectomy; or ii. Has had a bilateral oophorectomy, or iii. Has had a bilateral tubal ligation, or iv. Is post-menopausal (demonstrates total cessation of menses for greater than or equal to 1 year); OR
  2. Of childbearing potential, has a negative serum pregnancy test at screening, and agrees to one of the following contraceptives: i. An intrauterine device with a documented failure rate of less than 1% per year; ii. Vasectomized partner who is sterile prior to the subject's entry and is the sole sexual partner for that woman; iii. Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, during the clinical trial, and for at least 14 days after the last dose of investigational product; iv. Double barrier contraception defined as condom with spermicidal jelly, foam, suppository, or film; OR diaphragm with spermicide; OR male condom and diaphragm.

Exclusion Criteria:

* Brain metastases or spinal cord compression, unless treatment was completed at least 4 weeks before study entry, and stable without steroid treatment for at least 4 weeks.
* Evidence of severe or uncontrolled systemic diseases [e.g., unstable or uncompensated respiratory, cardiac (including life threatening arrhythmias)].
* Unresolved toxicity ≥ CTCAE Grade 2 from previous anti-cancer therapy except alopecia (if applicable) unless agreed that the patient can be entered after discussion with the Medical Monitor.
* Presence of cardiac impairment defined as:

  1. prior history of cardiovascular disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions; OR
  2. history of myocardial infarction/active ischemic heart disease within one year of study entry; OR
  3. uncontrolled dysrhythmias; OR
  4. poorly controlled angina
* Participation in a trial of an investigational agent within the prior 30 days
* Pregnant or breast-feeding.
* High volume peritoneal or pleural effusions requiring centesis more frequently than every 14 days.
* Poorly controlled or refractory (grade 3-4) hepatic encephalopathy.
* History of allogeneic stem cell or solid organ transplantation.
* Prior history of pneumonitis/interstitial lung disease.
* Receipt of live vaccine within 30 days.
* Active or prior documented autoimmune or inflammatory disorders (including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis). The following are exceptions to this criterion:

  1. Vitiligo or alopecia.
  2. Autoimmune-related hypothyroidism stable on thyroid replacement therapy.
  3. Any chronic skin condition that does not require systemic therapy.
  4. Controlled type 1 diabetes mellitus who are on an insulin regimen.
  5. Celiac disease controlled by diet alone.
  6. Without active disease in the last 5 year.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra-articular injection).
  2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
  3. Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
* Any concurrent condition that, in the investigator's opinion, makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  The primary endpoint is the number and frequency of adverse events related to cryoablation and hepatic artery infusion of SD-101 in combination with durvalumab and tremelimumab.
  Adverse events (AEs) during the 6 months following Cryo+SD-101 will be recorded. The NCI CTCAE version 5.0 will be used to grade adverse events. Incidence of AEs will be summarized by event type, grade and body system. Particularly, the rates of infusion reactions, major bleeding, major infection, and grade 3 or above non-infection adverse events will be reported. The proportion of patients having each type of adverse event will be summarized along with a corresponding 90% confidence interval calculated using the exact method. The rate and 90% exact CI of subjects who experience serious adverse events will also be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Burgoyne, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No